CLINICAL TRIAL: NCT00773682
Title: Efficacy and Tolerability of Mud Packs Therapy in Osteoarthritis of the Hands: a One Year Follow-up
Brief Title: Efficacy and Tolerability of Mud Packs Therapy in Osteoarthritis of the Hand
Acronym: mdph
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, medical doctor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 339/07
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2008-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; hands; mud-packs therapy; balneotherapy; Osteoarthritis of the hands
MeSH Terms: conditions — Osteoarthritis | interventions — Balneology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: local mud-pack therapy and balneotherapy — Patients will be treated with local mud-pack application on the hands for 20 minutes and thermal-mineral bath once a day for 15 days.

SUMMARY:
Objective

To assess both the short-term and the long term effectiveness of spa therapy in patients with primary hand osteoarthritis (OA) in a single blind, prospective controlled, randomized trial.

DETAILED DESCRIPTION:
Osteoarthritis is the most common form of joint disease and a major contributor of disability in older people. Current treatment of OA include pharmacological and non-pharmacological modalities. Spa therapy has a long history in the treatment of OA, but few articles have evaluated the effectiveness of thermal treatment in patients with primary OA of the hands.

The aim of this study is to assess the duration of the clinical effectiveness of mud-packs application and mineral bath in patients with primary OA of the hands in a single blind, controlled, randomized trial.

Our study will follow the patients for a longer period of time (12 months) than was done in previous studies.

60 outpatients will be enrolled; 30 patients will be treated with a combination of daily local mud packs and mineral bath water from the spa centre of Fonteverde Natural Spa Resort (San Casciano Terme, Siena, Italy) for two weeks; 30 patients will continue regular, routine ambulatory care. Patients will be assessed at baseline time, after 2 weeks, after 3, 6, 9 and 12 months following the beginning of the study and will be evaluated by VAS for spontaneous pain, Dreiser Algofunctional index, HAQ, AIMS1 and symptomatic drugs consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from osteoarthritis of the hands according to the ACR criteria

Exclusion Criteria:

* Patients suffering from any other rheumatological disease other than osteoarthritis
* Patients that have been treated with mud-pack therapy and balneotherapy in the last 9 months
* Contraindications to mud-packs and balneotherapy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Algofunctional state and quality of life | two weeks, three , six, nine and twelve months

SECONDARY OUTCOMES:
Consumption of symptomatic drugs and tolerability | two weeks, three, six, nine and twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Fioravanti, md, Principal Investigator — Rheumatology Unit- Azienda Ospedaliera Universitaria Senese-siena
Locations (1):
- Rheumatology Unit Azienda Ospedaliera Universitaria Senese, Siena, Siena, Italy

REFERENCES:
- [Background] Fioravanti A, Perpignano G, Tirri G, Cardinale G, Gianniti C, Lanza CE, Loi A, Tirri E, Sfriso P, Cozzi F. Effects of mud-bath treatment on fibromyalgia patients: a randomized clinical trial. Rheumatol Int. 2007 Oct;27(12):1157-61. doi: 10.1007/s00296-007-0358-x. Epub 2007 May 23. PMID 17520260
- [Background] Cantarini L, Leo G, Giannitti C, Cevenini G, Barberini P, Fioravanti A. Therapeutic effect of spa therapy and short wave therapy in knee osteoarthritis: a randomized, single blind, controlled trial. Rheumatol Int. 2007 Apr;27(6):523-9. doi: 10.1007/s00296-006-0266-5. Epub 2006 Nov 15. PMID 17106661
- [Background] Fioravanti A, Valenti M, Altobelli E, Di Orio F, Nappi G, Crisanti A, Cantarini L, Marcolongo R. Clinical efficacy and cost-effectiveness evidence of spa therapy in osteoarthritis. The results of "Naiade" Italian Project. Panminerva Med. 2003 Sep;45(3):211-7. PMID 14618120